CLINICAL TRIAL: NCT02665377
Title: Prevention of Akute Kidney Injury With Human Atrial Natriuretic Peptide in Patients Undergoing Heart Transplant.
Brief Title: Prevention of Akute Kidney Injury, Hearttransplant, ANP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Maria Tholén, MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SahlgrenskaUHMT01
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Atrial Natriuretic Factor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ANP (Active Comparator): Infusion of h-ANP at dose of 50ng/kg/min fore 5 days, starting at the induction of anesthesia.
  Interventions: Drug: ANP
- Placebo (Placebo Comparator): Infusion of NaCl at the same volyme as for ANP for 5 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANP
  Arms: ANP
Drug: Placebo
  Arms: Placebo

SUMMARY:
Prospective, blinded, placebo-controlled trial. Patients: Adult patients (>18 years of age) undergoing de novo Htx, with a preoperative GFR > 30ml/min, not receiving an ABO-incompatible organ with an ischemia time of > 6 hours. A donor age > 70 years is an exclusion criteria.

Intervention: Infusion of h-ANP fore five days, starting at the induction of anesthesia.

Outcome: Kidney function, evaluated with serum creatinine day 1-7 and kidney clearance, 4-5 Days after Htx plus after 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* De novo Htx.
* Preoperative GFR > 30ml/min/1,73m2.
* >18 years old.
* Written consent.

Exclusion Criteria:

* Multi organ transplantation or previous heart transplant.
* ECMO
* Donor age > 70 years.
* Dialysis.
* ABO-incompatible organ.
* Donor heart ischemia time > 6 tim.
* Known kidney disease.
* Other planed study within 2 mounth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-09-25 (Actual); Primary Completion 2022-01-08 (Actual); Study Completion 2022-01-08 (Actual)

PRIMARY OUTCOMES:
GFR 4-5 days after Htx | 4-5 days

SECONDARY OUTCOMES:
GFR 1 year after Htx | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Erik Ricksten, Prof, Principal Investigator — Sahlgrenska universitetssjukhuset
Locations (1):
- Sahlgrenska sjukhuset, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hashimoto H, Yamada H, Murata M, Watanabe N. Diuretics for preventing and treating acute kidney injury. Cochrane Database Syst Rev. 2025 Jan 29;1(1):CD014937. doi: 10.1002/14651858.CD014937.pub2. PMID 39878152